CLINICAL TRIAL: NCT04593407
Title: Endoscopic Mucosal Resection Versus Endoscopic Submucosal Dissection for Laterally Spreading Lesions Non Granular-Flat Elevated Type (LSL-NG-FE) ≥ 20 mm and LSLs-Granular Mixed Type ≥ 30 mm. A Randomized, Non-inferiority Trial.
Brief Title: Endoscopic Mucosal Resection Versus Endoscopic Submucosal Dissection for Colorectal Laterally Spreading Lesions.
Acronym: intERsection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: José Carlos Marín Gabriel (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other)
Responsible Party: Sponsor-Investigator, José Carlos Marín Gabriel, Principal Investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: intERsection-19/281
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms, Colorectal
Keywords: Colonic Polyps; large laterally spreading lesion; colonic adenoma; Endoscopic submucosal dissection; Endoscopic Mucosal Resection; Adenoma; Polyps; Pathological Conditions, Anatomical; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Intestinal Polyps
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Adenoma; Polyps; Pathological Conditions, Anatomical; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Intestinal Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Mucosal Resection (EMR): (Active Comparator): Piecemeal EMR is a conventional endoscopic resection technique. A submucosal injection of a large volume of a solution (normal saline or other) with or without dilute epinephrine (1/10,000) with or without indigo carmine is performed. Then, sequential piecemeal resection is performed with use of a combination of stiff-type snares. At the end of the procedure when macroscopically visible adenoma has been totally resected, a snare tip soft coagulation (STSC) of the margin of the scar is performed to eliminate non visible residual neoplastic tissue. This procedure is quicker and safer than ESD but led to more recurrent disease (around 20% with the standard technique but recently reduced to 5% after the introduction of STSC)
  Interventions: Procedure: Endoscopic mucosal resection (EMR)
- : Endoscopic Submucosal Dissection (ESD): (Experimental): ESD is a newer resection technique that allows en bloc resection for large LSLs. A submucosal injection is also needed but, in this case, different endo-knives are used to achieve the resection instead of diathermic snares. The en bloc resection allows a more precise pathological analysis and the risk of recurrence is lower (<2%) when margins are tumor-free.
  Interventions: Procedure: Endoscopic submucosal dissection (ESD)

INTERVENTIONS:
Procedure: Endoscopic mucosal resection (EMR) — Endoscopic mucosal resection (EMR) is an endoscopic resection technique that allows the removal of large colorectal lesions using a conventional "lift-and-cut" procedure or an underwater technique
  Arms: Endoscopic Mucosal Resection (EMR):
Procedure: Endoscopic submucosal dissection (ESD) — Endoscopic submucosal dissection (ESD) is an endoscopic procedure that allows dissection of larger colorectal lesions in one piece using endoknives.
  The procedure is technically more difficult, much more time-consuming than EMR, mandates multiday hospital admission and has an increased risk of perforation.
  Arms: : Endoscopic Submucosal Dissection (ESD):

SUMMARY:
EMR and ESD are both effective and safe and are associated with a very low risk of procedure related mortality when performed for colorectal laterally spreading lesions (LSL).

Some kind of LSLs have a low risk of submucosal invasive carcinoma (SMIC) or these foci are found in well demarcated areas of the tumor. This is the case of the non-granular flat elevated (LSN-NG-FE) and the LSLs-G mixed subtypes.

The investigators aim to assess if piecemeal EMR (the older technique) for LSLs-G mixed type > 30 mm and LSLs-NG FE type > 20 mm is not inferior to ESD (the new treatment) for the need of additional surgery in the mid-term.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is curative for lesions with superficial submucosal invasive carcinoma (s-SMIC) and favourable histological features. The procedure is performed mainly for laterally spreading lesions (LSLs) and is the reference treatment for these neoplasms in Asian countries nowadays. LSLs can be granular (G) or non-granular (NG). Most LSLs-G homogenous type are superficial and can be resected by EMR because SMIC is often lacking. On the other hand, since LSLs-G mixed type > 20 - 30 mm have a higher prevalence of SMIC when compared with the homogenous subtype, Asian experts now recommend ESD for this kind of tumors. However, some years ago, EMR had been suggested for LSLs-G mixed type if the largest nodule was resected first and the histological assessment was done separately. The rationale for the latter approach is that the invasive component is usually found within the large nodule.

Conversely, the prevalence of SMIC is higher in LSLs-NG PD type, therefore, ESD is the preferred therapeutic intervention. In addition, LSLs-NG FE type have been associated with multifocal invasion in Japanese studies. However, in Western countries, the percentage of SMIC in LSLs-NG FE type > 20 mm seems much lower than previously described in Asian series. Thus, the investigators do not know if EMR might be enough to remove these tumours.

Furthermore, if the risk of s-SMIC is low, the recurrence rates for ESD in these kind of lesions (LSL-G mixed type > 30 mm and LSL-NG FE type > 20 mm) might be comparable to that of piecemeal EMR, in terms of curative resection (avoiding the need for surgery) in the mid-term. When performing an EMR, recurrences are more frequent, but they are largely inconsequential because it is usually unifocal, diminutive and easily can be managed endoscopically on subsequent sessions.

In order to clarify the controversial issue of performing colorectal ESD in Western countries, the investigators aim to assess if piecemeal EMR (the older technique) for LSLs-G mixed type > 30 mm and LSLs-NG FE type > 20 mm is not inferior to ESD (the new treatment) for the need of additional surgery in the mid-term.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years old).
* LSL-NG FE type ≥ 20mm or LST-G mixed type ≥30mm who have not been previously treated or received submucosal injection, regardless of their location in the colon.
* LSL-NG FE type ≥ 20mm or LST-G mixed type ≥30mm WITHOUT a demarcated area
* The patient must have undergone a complete colonoscopy, reaching the cecum, to detect possible synchronous lesion. If this procedure has not been done previously, it will be performed prior to the inclusion of the patient in the study.
* Patients able to fill in questionnaires written in Spanish or English.

Exclusion Criteria:

* Contra-indication to colonoscopy.
* Contra-indication to general anesthesia.
* Inability to stop antiplatelet agents and anti-coagulant according to the European Society of Gastro-Intestinal Endoscopy guidelines.
* Patients with > 1 lesion meeting the inclusion criteria.
* LSL-NG FE type ≥ 20mm or LST-G ≥30mm mixed type that have been previously treated (Recurrence or residual lesion after previous endoscopic or surgical treatment).
* LSL-NG FE type ≥ 20mm or LST-G ≥30mm mixed type with previous submucosal injection, even if a resection attempt with a snare was not finally performed.
* Lesions with suspicion of deep submucosal invasive carcinoma: depression or invasive pit-pattern (Vi within a demarcated area or Vn).
* Submucosal mass like elevation within a LSL-NG FE type.
* LSLs having a previous biopsy or tattooing. Previous biopsies of the lesion should only be allowed if LSL-G mixed type > 30 mm and samples were taken out of the flat area.
* LSL-G with a Buddha like deformation (Polyp on polyp)
* LSL involving a surgical anastomosis.
* LSL involving the appendicular orifice.
* LSL involving the terminal ileum.
* Patient's refusal to participate in the study
* Presence of inflammatory bowel disease
* Pregnant or lactating women.
* Hereditary colorectal cancer syndrome or hereditary polyposis.
* Patient under legal protection and or deprived of liberty by judicial or administrative decision.
* Patient already participating in an interventional clinical research protocol
* Patient who cannot be followed for the duration of the study.
* Inability to sign the informed consent of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of surgical referral after treatment | Month 18
  Compare between two groups.

SECONDARY OUTCOMES:
En bloc resection rate | Month 1
  Compare between two groups
R0 resection rate | Month 1
  Compare between two groups
Duration of the procedure | Month 1
  Compare between two groups
Percentage of curative resection rates without surgery | Month 18
  Compare between two groups
Proportion of cases in which the endoscopist has to change technique to the alternative procedure | Month 1
  Compare between two groups
Cumulative complications rate after treatment | Month 1 and 18
  Compare between two groups

CONTACTS AND LOCATIONS:
Overall Officials: José C. Marín-Gabriel, Assoc. Prof., Study Director — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario "12 de Octubre", Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgess NG, Hourigan LF, Zanati SA, Brown GJ, Singh R, Williams SJ, Raftopoulos SC, Ormonde D, Moss A, Byth K, Mahajan H, McLeod D, Bourke MJ. Risk Stratification for Covert Invasive Cancer Among Patients Referred for Colonic Endoscopic Mucosal Resection: A Large Multicenter Cohort. Gastroenterology. 2017 Sep;153(3):732-742.e1. doi: 10.1053/j.gastro.2017.05.047. Epub 2017 Jun 2. PMID 28583826
- [Background] Uraoka T, Saito Y, Matsuda T, Ikehara H, Gotoda T, Saito D, Fujii T. Endoscopic indications for endoscopic mucosal resection of laterally spreading tumours in the colorectum. Gut. 2006 Nov;55(11):1592-7. doi: 10.1136/gut.2005.087452. Epub 2006 May 8. PMID 16682427
- [Background] Moss A, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Burgess NG, Sonson R, Byth K, Bourke MJ. Long-term adenoma recurrence following wide-field endoscopic mucosal resection (WF-EMR) for advanced colonic mucosal neoplasia is infrequent: results and risk factors in 1000 cases from the Australian Colonic EMR (ACE) study. Gut. 2015 Jan;64(1):57-65. doi: 10.1136/gutjnl-2013-305516. Epub 2014 Jul 1. PMID 24986245
- [Background] Albeniz E, Pellise M, Gimeno-Garcia AZ, Lucendo AJ, Alonso-Aguirre PA, Herreros de Tejada A, Alvarez MA, Fraile M, Herraiz Bayod M, Lopez Roses L, Martinez Ares D, Ono A, Parra Blanco A, Redondo E, Sanchez-Yague A, Soto S, Diaz-Tasende J, Montes Diaz M, Rodriguez-Tellez M, Garcia O, Zuniga Ripa A, Hernandez Conde M, Alberca de Las Parras F, Gargallo CJ, Saperas E, Munoz Navas M, Gordillo J, Ramos Zabala F, Echevarria JM, Bustamante M, Gonzalez-Haba M, Gonzalez-Huix F, Gonzalez-Suarez B, Vila Costas JJ, Guarner Argente C, Mugica F, Cobian J, Rodriguez Sanchez J, Lopez Viedma B, Pin N, Marin Gabriel JC, Nogales O, de la Pena J, Navajas Leon FJ, Leon Brito H, Remedios D, Esteban JM, Barquero D, Martinez Cara JG, Martinez Alcala F, Fernandez-Urien I, Valdivielso E. Clinical guidelines for endoscopic mucosal resection of non-pedunculated colorectal lesions. Rev Esp Enferm Dig. 2018 Mar;110(3):179-194. doi: 10.17235/reed.2018.5086/2017. PMID 29421912
- [Background] Yang D, Othman M, Draganov PV. Endoscopic Mucosal Resection vs Endoscopic Submucosal Dissection For Barrett's Esophagus and Colorectal Neoplasia. Clin Gastroenterol Hepatol. 2019 May;17(6):1019-1028. doi: 10.1016/j.cgh.2018.09.030. Epub 2018 Sep 26. PMID 30267866
- [Background] Fujiya M, Tanaka K, Dokoshi T, Tominaga M, Ueno N, Inaba Y, Ito T, Moriichi K, Kohgo Y. Efficacy and adverse events of EMR and endoscopic submucosal dissection for the treatment of colon neoplasms: a meta-analysis of studies comparing EMR and endoscopic submucosal dissection. Gastrointest Endosc. 2015 Mar;81(3):583-95. doi: 10.1016/j.gie.2014.07.034. Epub 2015 Jan 13. PMID 25592748
- [Background] Arezzo A, Passera R, Marchese N, Galloro G, Manta R, Cirocchi R. Systematic review and meta-analysis of endoscopic submucosal dissection vs endoscopic mucosal resection for colorectal lesions. United European Gastroenterol J. 2016 Feb;4(1):18-29. doi: 10.1177/2050640615585470. Epub 2015 May 5. PMID 26966519
- [Background] Moss A, Bourke MJ, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Chen RY, Byth K. Endoscopic mucosal resection outcomes and prediction of submucosal cancer from advanced colonic mucosal neoplasia. Gastroenterology. 2011 Jun;140(7):1909-18. doi: 10.1053/j.gastro.2011.02.062. Epub 2011 Mar 8. PMID 21392504
- [Background] Wang J, Zhang XH, Ge J, Yang CM, Liu JY, Zhao SL. Endoscopic submucosal dissection vs endoscopic mucosal resection for colorectal tumors: a meta-analysis. World J Gastroenterol. 2014 Jul 7;20(25):8282-7. doi: 10.3748/wjg.v20.i25.8282. PMID 25009404
- [Background] Belderbos TD, Leenders M, Moons LM, Siersema PD. Local recurrence after endoscopic mucosal resection of nonpedunculated colorectal lesions: systematic review and meta-analysis. Endoscopy. 2014 May;46(5):388-402. doi: 10.1055/s-0034-1364970. Epub 2014 Mar 26. PMID 24671869
- [Background] Uraoka T, Parra-Blanco A, Yahagi N. Colorectal endoscopic submucosal dissection in Japan and Western countries. Dig Endosc. 2012 May;24 Suppl 1:80-3. doi: 10.1111/j.1443-1661.2012.01279.x. PMID 22533758
- [Background] Oyama T, Yahagi N, Ponchon T, Kiesslich T, Berr F. How to establish endoscopic submucosal dissection in Western countries. World J Gastroenterol. 2015 Oct 28;21(40):11209-20. doi: 10.3748/wjg.v21.i40.11209. PMID 26523097
- [Background] Repici A, Hassan C, De Paula Pessoa D, Pagano N, Arezzo A, Zullo A, Lorenzetti R, Marmo R. Efficacy and safety of endoscopic submucosal dissection for colorectal neoplasia: a systematic review. Endoscopy. 2012 Feb;44(2):137-50. doi: 10.1055/s-0031-1291448. Epub 2012 Jan 23. PMID 22271024
- [Background] Emmanuel A, Gulati S, Burt M, Hayee B, Haji A. Colorectal endoscopic submucosal dissection: patient selection and special considerations. Clin Exp Gastroenterol. 2017 Jul 13;10:121-131. doi: 10.2147/CEG.S120395. eCollection 2017. PMID 28761366
- [Background] Oka S, Tanaka S, Kanao H, Oba S, Chayama K. Therapeutic strategy for colorectal laterally spreading tumor. Dig Endosc. 2009 Jul;21 Suppl 1:S43-6. doi: 10.1111/j.1443-1661.2009.00869.x. PMID 19691733
- [Background] Saito Y, Uraoka T, Yamaguchi Y, Hotta K, Sakamoto N, Ikematsu H, Fukuzawa M, Kobayashi N, Nasu J, Michida T, Yoshida S, Ikehara H, Otake Y, Nakajima T, Matsuda T, Saito D. A prospective, multicenter study of 1111 colorectal endoscopic submucosal dissections (with video). Gastrointest Endosc. 2010 Dec;72(6):1217-25. doi: 10.1016/j.gie.2010.08.004. Epub 2010 Oct 27. PMID 21030017
- [Background] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Background] Russo P, Barbeiro S, Awadie H, Libanio D, Dinis-Ribeiro M, Bourke M. Management of colorectal laterally spreading tumors: a systematic review and meta-analysis. Endosc Int Open. 2019 Feb;7(2):E239-E259. doi: 10.1055/a-0732-487. Epub 2019 Jan 30. PMID 30705959
- [Background] Bourke MJ, Neuhaus H, Bergman JJ. Endoscopic Submucosal Dissection: Indications and Application in Western Endoscopy Practice. Gastroenterology. 2018 May;154(7):1887-1900.e5. doi: 10.1053/j.gastro.2018.01.068. Epub 2018 Mar 2. PMID 29486200
- [Background] Thoguluva Chandrasekar V, Spadaccini M, Aziz M, Maselli R, Hassan S, Fuccio L, Duvvuri A, Frazzoni L, Desai M, Fugazza A, Jegadeesan R, Colombo M, Dasari CS, Hassan C, Sharma P, Repici A. Cold snare endoscopic resection of nonpedunculated colorectal polyps larger than 10 mm: a systematic review and pooled-analysis. Gastrointest Endosc. 2019 May;89(5):929-936.e3. doi: 10.1016/j.gie.2018.12.022. Epub 2019 Jan 9. PMID 30639542
- [Background] Bahin FF, Heitman SJ, Rasouli KN, Mahajan H, McLeod D, Lee EYT, Williams SJ, Bourke MJ. Wide-field endoscopic mucosal resection versus endoscopic submucosal dissection for laterally spreading colorectal lesions: a cost-effectiveness analysis. Gut. 2018 Nov;67(11):1965-1973. doi: 10.1136/gutjnl-2017-313823. Epub 2017 Oct 7. PMID 28988198
- [Background] Yamada M, Saito Y, Sakamoto T, Nakajima T, Kushima R, Parra-Blanco A, Matsuda T. Endoscopic predictors of deep submucosal invasion in colorectal laterally spreading tumors. Endoscopy. 2016 May;48(5):456-64. doi: 10.1055/s-0042-100453. Epub 2016 Feb 26. PMID 26919264
- [Background] Bogie RMM, Veldman MHJ, Snijders LARS, Winkens B, Kaltenbach T, Masclee AAM, Matsuda T, Rondagh EJA, Soetikno R, Tanaka S, Chiu HM, Sanduleanu-Dascalescu S. Endoscopic subtypes of colorectal laterally spreading tumors (LSTs) and the risk of submucosal invasion: a meta-analysis. Endoscopy. 2018 Mar;50(3):263-282. doi: 10.1055/s-0043-121144. Epub 2017 Nov 27. PMID 29179230
- [Background] Tate DJ, Awadie H, Bahin FF, Desomer L, Lee R, Heitman SJ, Goodrick K, Bourke MJ. Wide-field piecemeal cold snare polypectomy of large sessile serrated polyps without a submucosal injection is safe. Endoscopy. 2018 Mar;50(3):248-252. doi: 10.1055/s-0043-121219. Epub 2017 Nov 23. PMID 29169195
- [Background] Gupta S, Miskovic D, Bhandari P, Dolwani S, McKaig B, Pullan R, Rembacken B, Riley S, Rutter MD, Suzuki N, Tsiamoulos Z, Valori R, Vance ME, Faiz OD, Saunders BP, Thomas-Gibson S. A novel method for determining the difficulty of colonoscopic polypectomy. Frontline Gastroenterol. 2013 Oct;4(4):244-248. doi: 10.1136/flgastro-2013-100331. Epub 2013 Jun 1. PMID 28839733
- [Background] Klein A, Tate DJ, Jayasekeran V, Hourigan L, Singh R, Brown G, Bahin FF, Burgess N, Williams SJ, Lee E, Sidhu M, Byth K, Bourke MJ. Thermal Ablation of Mucosal Defect Margins Reduces Adenoma Recurrence After Colonic Endoscopic Mucosal Resection. Gastroenterology. 2019 Feb;156(3):604-613.e3. doi: 10.1053/j.gastro.2018.10.003. Epub 2018 Oct 6. PMID 30296436